CLINICAL TRIAL: NCT05494424
Title: Cognitive Rehabilitation in Post-COVID-19 Condition: A Study Protocol for a Randomized Controlled Trial
Brief Title: Cognitive Rehabilitation in Post-COVID-19 Condition
Acronym: TRAINCOVID
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: University of Oslo (Other); Icahn School of Medicine at Mount Sinai (Other); University of Toronto (Other); UiT The Arctic University of Norway (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Traincovid
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
Keywords: Rehabilitation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Goal Management Training (GMT) (Experimental): Internet-delivered group-based GMT to groups of six participants in six two-hour sessions delivered weekly (five weeks). Manualized intervention.
  Interventions: Behavioral: Goal Management Training (GMT)
- Wait list (No Intervention): Wait list control condition

INTERVENTIONS:
Behavioral: Goal Management Training (GMT) — Goal Management Training is a cognitive rehabilitation intervention that relies on metacognitive strategies to reengage top-down attention processes, in addition to teaching problem-solving techniques, attempting to address executive dysfunctions.
  Other Names: GMT
  Arms: Goal Management Training (GMT)

SUMMARY:
Post-COVID-19 condition is frequently comprised of persistent cognitive sequela, including deficits in attention and executive functions (EFs). Goal Management Training (GMT) is a cognitive rehabilitation (CR) intervention for improving attention and EFs that has received empirical support in studies of other patient groups. The present study aims to determine the efficacy of GMT for improving everyday attention and EFs in adults who experience persistent cognitive deficits after COVID-19. The study is a randomized controlled trial (RCT), comparing the efficacy of GMT to a wait list control condition (WL), for improving persistent cognitive sequela in post-COVID-19 condition. The study aims to recruit 120 participants aged 18 to 65 years with a history of laboratory- or home-test confirmed, SARS-CoV-2 infection and perceived attentional and EF difficulties in daily life that have lasted for at least two months and that cannot be explained by an alternative diagnosis. Participants will be randomized to either group-based GMT (n = 60) or WL (n = 60). GMT will be internet-delivered to groups of six participants in six two-hour sessions delivered weekly (five weeks). The primary outcome will be the Metacognition Index of the Behavior Rating Inventory of Executive Function - Adult Version, a self-report measure assessing everyday EF difficulties, at six months post-treatment. Secondary outcomes include performance-based neurocognitive measures and rating scales of cognition, emotional health, quality of life, and fatigue.

Secondary aims include to explore to what extent potential early change predicts outcome, and to examine what characterize those who profit from GMT, in addition to describe the neurocognitive and emotional health in a Covid-19 sample. The investigators will also examine potential effects of GMT at 2- and 5-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* history of laboratory- or home-test confirmed, SARS-CoV-2 infection
* perceived cognitive difficulties (attention, memory, EF) affecting everyday functioning that have lasted for at least two months and that cannot be explained by an alternative diagnosis
* age between 18-65 years

Exclusion Criteria:

* ongoing alcohol- or substance abuse, premorbid insult and/or comorbid neurological disease, severe neurocognitive problems interfering with the capacity to participate, sensory disorders biasing cognitive assessment, psychotic disorders, lack of proficiency in Norwegian, and being previously enrolled in a GMT trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
The Metacognition Index from the Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A) | Change from baseline up to 6 months
  Self-report measure of daily life executive function (metacognition). Range:70-210. Higher score indicate greater executive dysfunction.

SECONDARY OUTCOMES:
The Behaviour regulation Index from Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A) | Change from baseline up to 6 months
  Self-report measure of daily life executive function (behaviour regulation). Range: 70-210. Higher score indicate greater executive dysfunction.
Cambridge Neuropsychological Test Automated Battery (CANTAB), subtests: Spatial Working Memory, Rapid Visual Information Processing, One Touch Stockings of Cambridge | Change from baseline up to 6 months
  Performance-based neurocognitive test battery
The Hospital Anxiety and Depression Scale | Change from baseline up to 6 months
  Self-report measure of symptoms of anxiety and depression. The maximum score is 21 for depression and 21 for anxiety, range 0-21 on each scale. A higher score = more symptoms.
The Generalized Self-Efficacy Scale | Change from baseline up to 6 months
  Self-report measure of self-efficacy. Range:10-40. Higher score indicate higher self-efficacy.
Fatigue Severity Scale | Change from baseline up to 6 months
  Self-report measure of fatigue. 7 items. Range 7-49. Higher score indicate more fatigue.
The Perceived Deficits Questionnaire | Change from baseline up to 6 months
  Self-report measure of daily-life cognitive difficulties. The total score range from 0 to 80, with a higher score indicating greater perceived cognitive impairment.
Everyday Memory Questionnaire | Change from baseline up to 6 months
  Self-report measure of daily-life cognitive difficulties. The total score range from 0 to 52, with a higher score indicating greater perceived cognitive impairment.
RAND 12-Item Health Survey (RAND-12) | Change from baseline up to 6 months
  Self-report measure of quality of life. Range 0-10; a high score defines a more favorable health state.
EuroQol five-dimension scale questionnaire (EQ-5D) | Change from baseline up to 6 months
  Self-report measure of quality of life. The range of the EQ-5D index scores is 0 to 1 (1 indicates the best health state), but negative scores as low as-0.59 are possible for health states deemed to be worse than death.
DePaul Symptom Questionnaire short version | Change from baseline up to 6 months
  Self-report measure of fatigue symptoms. 14 items. The total score range from 0 to 56 for both frequency and severity for each item.
Insomnia Severity Index | Change from baseline up to 6 months
  Self-report measure of insomnia. Range: 0-28. Higher score indicate more acute symptoms of insomnia

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stubberud, PhD, Principal Investigator — University of Oslo and Lovisenberg Hospital
Locations (1):
- Lovisenberg Diaconal Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hagen BI, Lerdal A, Soraas A, Landro NI, Bo R, Smastuen MC, Becker J, Stubberud J. Cognitive rehabilitation in post-COVID-19 condition: A study protocol for a randomized controlled trial. Contemp Clin Trials. 2022 Nov;122:106955. doi: 10.1016/j.cct.2022.106955. Epub 2022 Oct 5. PMID 36208718